CLINICAL TRIAL: NCT01533311
Title: Prevalence and Characteristics of Nonpolypoid Colorectal Neoplasms - A Chinese Cohort Study
Status: Completed | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaobo Li, Shanghai Institute of Digestive Disease，Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai Jiao Tong University School of Medicine
Other Study IDs: rjxhnk03
Record Dates: First submitted 2012-02-11; First posted 2012-02-15 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Nonpolypoid Colorectal Neoplasms(NP-CRN)
Keywords: nonpolypoid colorectal neoplasms(NP-CRN); prevalence; histology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — All the lesions will be removed endoscopically or surgically and examined histologically by an independent gastrointestinal pathologist.
  Histological diagnosis is determined according to the World Health Organization (WHO) criteria.Pedunculated lesions are categorized according to Haggitt's classification.
Oversight: Data Monitoring Committee: No

SUMMARY:
The nonpolypoid colorectal neoplasms (NP-CRNs) are relatively common in patients with gastrointestinal alarm systoms. The depressed lesions have a greater risk of having cancer than flat and polypoid lesions.

ELIGIBILITY:
Inclusion Criteria:

* consecutive adult patients undergo colonoscopy by one endoscopist

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive adult patients undergo colonoscopy by one endoscopist from Jan 2009 to Dec 2010
Sampling Method: Non-Probability Sample
Enrollment: 1342 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)